CLINICAL TRIAL: NCT00602602
Title: A Phase II Study of Gemcitabine, Oxaliplatin and Bevacizumab Followed by 5-Fluorouracil, Oxaliplatin, Bevacizumab and Radiotherapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Bevacizumab, Combination Chemotherapy, and Radiation Therapy in Treating Patients Undergoing Surgery For Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000580812; UPCC-04206; GENENTECH-UPCC-04206; UPCC-805957
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Fluorouracil; Gemcitabine; Oxaliplatin; Immunohistochemistry; Endoscopic Mucosal Resection; Laparoscopy; Radiotherapy

ARMS (1):
- GemOx and Bev, then chemoradiation, then surgery (Experimental): Gemcitabine 1000 mg/m2 over 100 min on day 1 every 2 weeks
  Oxaliplatin 85 mg/m2 over 2 hours on day 2 every 2 weeks
  Bevacizumab 10 mg/kg over 90 minutes on day 1 every 2 weeks. Infusion duration may be shortened in subsequent courses if tolerated.
  One cycle is 2 weeks. Chemoradiation to begin prior to 4 weeks from last dose of Gem. Between 4 and 6 weeks following chemoradiotherapy, patients will undergo re-staging with CT or MRI and CA 19-9. If there is no evidence of disease progression, the patient will be referred to the surgeon for re-evaluation and consideration of surgical intervention
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: conventional surgery; Procedure: endoscopic biopsy; Procedure: laparoscopy; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: oxaliplatin
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: conventional surgery
Procedure: endoscopic biopsy
Procedure: laparoscopy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as gemcitabine, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab together with combination chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: The phase II trial is studying the side effects and how well giving bevacizumab together with gemcitabine, oxaliplatin, fluorouracil, and radiation therapy works in treating patients undergoing surgery for locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To describe the toxicity of bevacizumab with gemcitabine and oxaliplatin, when therapy is given before chemoradiotherapy, in patients with locally advanced pancreatic cancer.
* To describe the toxicity of bevacizumab with oxaliplatin, fluorouracil, and concomitant radiotherapy in these patients.
* To define progression-free survival, time to progression, and overall survival of patients treated with this regimen.

Second

* To determine the percentage of potentially resectable patients who are ultimately able to proceed to successful resection.
* To determine the relationship between markers of apoptosis in tumor cells (including MIF, CREB, HIF-1-alpha expression/polymorphism, and others) and response to therapy.
* To define response rates in patients treated with this regimen.

OUTLINE:

* Neoadjuvant therapy: Patients receive gemcitabine IV over 100 minutes and bevacizumab IV over 30-90 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Between 4-6 weeks after completion of initial therapy, patients undergo radiotherapy once daily, 5 days a week, for 5-6 weeks. Beginning within 48 hours after initiation of radiotherapy, patients receive fluorouracil IV continuously through completion of radiotherapy. Patients also receive concurrent oxaliplatin IV over 2 hours on days 1, 15 and 29 and bevacizumab IV on days 1 and 15.
* Surgery: Four to six weeks after completion of neoadjuvant therapy, patients undergo resection of the tumor. Patients with no evidence of disease progression and who undergo successful surgical intervention (i.e., R0 resection) proceed to adjuvant chemotherapy within the next 6-10 weeks.
* Adjuvant therapy: Patients receive gemcitabine and bevacizumab for 4 courses as in neoadjuvant therapy.

Patients undergo collection of tumor tissue samples at the time of diagnosis, prior to treatment by endoscopic ultrasound or laparoscopy, or during surgical resection following neoadjuvant therapy. Paraffin-embedded tumor tissue specimens obtained at baseline are analyzed by immunohistochemistry to assess tumor vascularity and angiogenic activity. Tumor vascularity is assessed via immunostaining of tumor specimens with the pan-endothelial cell marker, anti-CD34, for evaluation of tumor blood vessels. Angiogenic activity is assessed by analyzing pERK1/2, Ki67, and the pericyte coverage index in tumor specimens. Patients also undergo blood collection to determine plasma levels of VEGF at 4 weeks prior to initial chemotherapy and bevacizumab, at up to 48 hours prior to chemoradiotherapy and bevacizumab, and at up to 48 hours prior to adjuvant chemotherapy and bevacizumab.

After completion of study therapy, patients are followed every 2 months for the first year, and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Resectable, marginally resectable, or unresectable disease determined by one of the following:

    * Contrast-enhanced helical-CT scan
    * Endoscopic ultrasound with biopsy (in patients who do not have metastatic or grossly unresectable disease)
    * Dedicated pancreatic MRI
  * Tumor must be locally advanced or potentially resectable, as determined by one of the following:

    * Abutment of the portal or superior mesenteric veins, hepatic or superior mesenteric artery
    * Extension to the origin of gastroduodenal artery
    * Occlusion of the superior mesenteric vein for < 2 cm
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT

  * Marker elevation alone not allowed as justification for study entry
* Formalin-fixed, paraffin-embedded tumor tissue specimens from prior biopsy or surgical resection allowed for correlative studies
* No known brain metastases or tumor metastatic to the peritoneum, liver, or other organs

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥1,500/mm³
* Platelet count ≥ 100,000/mm³
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Bilirubin < 2.0 mg/dL (≤ 10 mg/dL for patients with biliary obstruction by tumor)

  * A biliary stent ≥ 9F or biliary bypass is required before treatment if there is biliary obstruction by tumor
* Urine protein:creatinine ratio ≤ 1.0
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant traumatic injury within the past 28 days
* No serious non-healing wounds, ulcers, or bone fractures
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No myocardial infarction, unstable angina, or cerebrovascular accident within the past 6 months
* No NYHA class II-IV congestive heart failure

  * Class II defined as symptoms of fatigue, dyspnea or other symptoms with ordinary physical activity
* No clinically significant peripheral vascular disease
* Pre-existing hypertension allowed, provided that the patient is receiving a stable antihypertensive regimen and has a blood pressure ≤ 150/100 mm Hg at the time of enrollment
* Must have adequate oral intake of > 1500 calories/day and be able to maintain hydration OR have access for supplemental enteral feeding (nasoenteral tube, feeding jejunostomy, or percutaneous endoscopic gastrostomy tube)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for pancreatic cancer
* More than 28 days since prior and no anticipated need for concurrent major surgical procedures
* More than 7 days since prior minor surgical procedures such as laparoscopy, fine needle aspirations, or core biopsies
* No treatment plan requiring treatment of > 50% of the liver at a dose > 30 Gy or > 50% of the total kidney volume at a dose > 18 Gy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No oral or parenteral anticoagulation unless patients is receiving a stable dose of anticoagulant

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Response rate pre-radiation chemotherapy and bevacizumab and after 5-6 weeks of concurrent chemoradiotherapy and bevacizumab | after 6-12 weeks
  Response rate pre-radiation chemotherapy and bevacizumab and after 5-6 weeks of concurrent chemoradiotherapy and bevacizumab
Progression-free survival | approximately 26 weeks
  to be assessed after completion of treatment

SECONDARY OUTCOMES:
Percentage of potentially resectable patients who are able to proceed to successful resection | approximately 12 weeks from initial chemo start
  after chemoradiation, those who can proceed to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States